CLINICAL TRIAL: NCT02185079
Title: The Effect of Metrics Based Performance Based Progression in Provision of Labor Epidural Analgesia on Clinical Performance and Clinical Outcome
Brief Title: The Effect of Metrics Based Performance Based Progression in Provision of Labor Epidural Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Karthikeyan Kallidaikurichi Srinivasan, Specialist Registrar,Anaesthetics,Cork University Hospital, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ECM4(i)06/05/2014
Record Dates: First submitted 2014-07-05; First posted 2014-07-09 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Labor Pain
Keywords: labor; epidural
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group C (Active Comparator): Conventional training for epidural catheter placement as per department protocols will be given to the trainees in this arm. Access to epidural simulator for 2 days will be given.
  Interventions: Behavioral: Conventional training
- Group M (Experimental): Conventional training for epidural catheter placement as per department protocols will be given to the trainees in this arm as well.Trainees in this arm in addition will be subjected to training to proficiency based on the metrics developed for labor epidural catheter placement in a epidural simulator.
  Interventions: Behavioral: Training to proficiency

INTERVENTIONS:
Behavioral: Training to proficiency — Conventional training for epidural catheter placement as per department protocols will be given to the trainees in this arm as well.Trainees in this arm in addition will be trained to proficience based on the metrics developed for labor epidural catheter placement in a epidural simulator.
  Arms: Group M
Behavioral: Conventional training — Conventional training for epidural catheter placement as per department protocols will be given to the trainees in this arm. Access to epidural simulator for 2 days will be given.
  Arms: Group C

SUMMARY:
Procedural skills are an important determinant of clinical outcomes for certain patient groups. Training for procedural skills in the medical profession is still largely based on an apprenticeship model. For example, trainees learning to perform epidural anaesthesia do so by "practicing" on patients under direct supervision by seniors (consultants or senior registrars/residents). Learning a complex and high risk procedural skill on patients is not ideal.

As medical training moves from apprentice based to competency based training along and as for the number of clinical learning opportunities for trainees is less, it is necessary to develop a comprehensive training programme which enables effective and efficient learning without compromising on patient safety. Metrics-based performance based progression has shown to improve clinical performance not only in novices but also in experts.

We envisage a standard methodology which could address the deficiencies in procedural training currently. This would entail development and validation of a set of metrics for a particular procedure, evaluation of a proficiency based progression training programme based on those metrics to and demonstration of improved clinical performance and clinical outcome associated with that programme. Although elements of this "end -end" approach have been demonstrated previously for various procedures, we propose to apply this methodology in its entirety to placement of a lumbar epidural catheter for analgesia for patients in labor. To date we have developed and are validating a set of metrics for this procedure. Proficiency based training leading to better procedural skills leading to better patient outcomes has not been studied so far. Epidural analgesia during labor lends itself as an excellent model for evaluating the whole process. It has a specific procedural skill which is closely linked to patient outcome which is measurable and occurs in finite time interval.

The hypothesis of the study is that in novice anaesthetic trainees, training with metrics based performance based progression in addition to improving the clinical performance will also reduce the failure rates of labor epidural analgesia to 5% when compared to 25% achieved by conventional training.

DETAILED DESCRIPTION:
This will be a prospective, randomized, double blind control study. Ethical committee approval and consent from both participating anaesthetist and patients will be obtained.

Trainees will be recruited from Cork University Hospital. Anaesthetic trainees with less than 2 years of experience in anaesthesia and who has performed less than 50 epidurals in the preceding 2 years (not limited to labor epidurals) will be requested to participate in the study.

The trainees will be randomized in to group 1 and group 2. In group 1, standardized conventional teaching and training for labor epidural analgesia will be used. In group 2, they will be trained by metrics based simulation to predetermined level of proficiency. Each trainee will then perform 10 labor epidural catheter insertions and the procedures will be video recorded with patients consent.

Observers blinded to the groups will be used for the data collection, outcome assessment and analysis. Failure rate of epidural will be assessed based on the occurrence of one or more of the following events,

1. Inadequate analgesia at 45 minutes from start of epidural needle placement.
2. Resiting epidural or abandoning the procedure.
3. Accidental Dural puncture.
4. Supervisor take over. The primary end point of the study is to compare difference in epidural failure rates between the two groups. Secondary end point will include assessment of clinical performance using metrics based assessment by two blinded reviewers based on video recordings and patient satisfaction with epidural analgesia. In addition to demographic data of the patients, duration of labor, cervical dilation at the time of insertion of the catheter, length of catheter inserted, time of insertion of catheter, experience of the operator and position of the patient during epidural placement will be noted. Age, sex and anaesthesia experience of the trainees will also be collected.

The estimated labor epidural failure rates for year 1 trainees is 25%.6 We hope to reduce the failure rate in interventional group to 5%. 48 procedures per group will be sufficient to show a statistically significant difference between the groups with p value of 0.05% and power of 80%. To allow for dropouts, 8 trainees per group will be recruited and each will perform 10 procedures making it a total of 80 procedures per group.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthetic trainees with less than 2 years of experience in anaesthesia and who has performed less than 50 epidurals in the preceding 2 years (not limited to labor epidurals) will be requested to participate in the study.

Exclusion Criteria:

* No tmeeting inclusion criteria
* Not consenting for study

Ages: 23 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Epidural failure rate | within 48 hours after completion of epidural
  Failure rate of epidural will be assessed based on the occurrence of one or more of the following events,
  1. Inadequate analgesia at 45 minutes from start of epidural needle placement.
  2. Resiting epidural or abandoning the procedure.
  3. Accidental Dural puncture.
  4. Supervisor take over.

SECONDARY OUTCOMES:
assessment of clinical performance using metrics based assessment | within 36 months after aquiring the video of epidrual catheter insertion procedure
  assessment of clinical performance using metrics based assessment will be done by two blinded reviewers based on video recordings
patient satisfaction with epidural analgesia | within 48 hours of completion of insertion of labor epidural catheter
  Patient will be asked to rate eidural as (a) satisfied, will want it again (b) Not satisfied - give reason in free text

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan Kallidaikurichi Srinivasan, FCARCSI,MD, Principal Investigator — Cork University Hospital
Locations (1):
- Cork University Hospital, Cork,Ireland, Cork, Ireland

REFERENCES:
- [Derived] Kallidaikurichi Srinivasan K, Gallagher A, O'Brien N, Sudir V, Barrett N, O'Connor R, Holt F, Lee P, O'Donnell B, Shorten G. Proficiency-based progression training: an 'end to end' model for decreasing error applied to achievement of effective epidural analgesia during labour: a randomised control study. BMJ Open. 2018 Oct 15;8(10):e020099. doi: 10.1136/bmjopen-2017-020099. PMID 30327396